CLINICAL TRIAL: NCT02751762
Title: A Prospective Investigation of the Risks of Opioid Misuse, Abuse, and Addiction Among Patients Treated With Opioids for the Treatment of Chronic Pain
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-1; Study 3033-1 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-04-06; First posted 2016-04-26 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples collected from consented study participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Longitudinal Cohort: Patients who have recently initiated long-term opioid therapy or initiated ER/LA opioid therapy
  Interventions: Other: Observation Only
- Cross-sectional Cohort: Patients who have been treated with opioids (including at least one ER/LA opioid) for greater than one year
  Interventions: Other: Observation Only

INTERVENTIONS:
Other: Observation Only — No Intervention

SUMMARY:
The purpose of this study is to quantify the serious risks of prescription opioid misuse or abuse or opioid use disorder (OUD) associated with the long term use of opioid analgesics for management of chronic pain, among patients prescribed opioid products.

DETAILED DESCRIPTION:
The Food and Drug Administration (FDA) has asked the companies that are New Drug Application (NDA) holders of extended-release/long-acting (ER/LA) opioids to conduct one or more studies to provide quantitative estimates of the serious risks of prescription opioid misuse or abuse or opioid use disorder associated with long-term use of opioid analgesics for management of chronic pain, among patients prescribed opioid products. Although abuse and misuse of prescription opioids have increased over the past decade, there is debate about the magnitude of misuse, abuse, and addiction among patients who are treated with prescription opioids for chronic pain. Further, although there appears to be comorbidity of opioid use disorders with other substance use and psychiatric disorders, there is insufficient data to estimate how the risk of these outcomes varies by the presence of risk factors among patients treated with opioids long-term. This study seeks to fill that gap. The primary objective is to quantify the serious risks of prescription opioid misuse or abuse or OUD associated with long-term use of opioid analgesics for management of chronic pain among patients prescribed opioid products. Patients will be recruited from seven Health Care System Research Network (HCSRN) sites; one U.S. Department of Veterans Affairs (VA) site; and clinics participating in two Primary Care Practice-Based Research Network sites. The data sources for the proposed study will be: 1) patient reported outcomes through in-person interviews (or phone if unavailable to participate in-person), 2) web-based assessments (or phone if unable to complete via web), and 3) electronic medical record and claims data. The study design includes two components: 1) a prospective longitudinal study of patients who have recently initiated long-term opioid therapy or initiated ER/LA opioid therapy, and 2) a cross-sectional study of patients who have been treated with opioids (including at least one ER/LA opioid) for at least one year.

ELIGIBILITY:
Eligibility Criteria for the Prospective Study

Inclusion Criteria:

* Initiation* of ER/LA opioid therapy that includes 28+ days of an ER/LA followed by a subsequent ER/LA prescription (ER/LA initiators) or initiation** of long-term opioid therapy (LtOT - 90+ days of use) with ER/LA and/or Schedule II IR/SA opioids (LtOT initiators).
* Age 18-79 years at incident prescription
* Enrolled in the health plan (HCSRN sites) or regularly receiving care in the health system (VA and PBRNs) for at least 12 months prior to incident use of opioids
* Ability to complete interview/self-administered questionnaires in English
* Willing and able to provide informed consent

  * Initiation or new use of ER/LA therapy defined as no ER/LA opioid use in the prior six-months ** Initiation or new LtOT use defined as no ER/LA or Schedule II IR/SA opioid use in the prior six-months

Exclusion Criteria:

* Not using an ER/LA or Schedule II IR/SA opioid at the time of recruitment or first interview (self-report)
* Cognitive impairment that interferes with the ability to consent or participate in the interview
* Unavailable for 12 months of follow-up (self-report)
* Receiving hospice care (EHR and recruitment screening)
* Diagnosis of a terminal illness in the prior 12 months per chart review or recruitment screening
* Existing opioid use disorder (ICD-9 and ICD-10 diagnosis codes)
* Medication assisted treatment with methadone or buprenorphine (self-report)

Eligibility Criteria - Cross Sectional Study:

Inclusion Criteria:

* Regular opioid use in the past year with at least 1 prescription for an ER/LA opioid. See Figure 4 for specifics on how these criteria are operationalized.
* Age 18-79 years at index prescription Enrolled in the health plan (HCSRN sites) or regularly receiving care in the health system (VA and PBRNs) for at least 12 months prior to index date.
* Ability to complete interview/self-administered questionnaires in English
* Willing and able to provide informed consent

Exclusion Criteria:

* Not using an opioid at the time of recruitment or first interview (self-report)
* Cognitive impairment that interferes with the ability to consent or participate in the interview
* Receiving hospice care (EHR and recruitment screening)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Of the approximately 2300 eligible subjects in the prospective study, approximately 2200 will be from the HCSRN sites, 25 from the VA, and a total of 100 from the PBRN sites. Sampling and recruitment strategies for the cross-sectional study will parallel those used to identify the prospective sample.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Prospective Longitudinal study: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ) | Change from baseline at up to one year
  Estimation of the incidence of misuse and abuse associated with long-term use of opioids for chronic pain.
Prospective Longitudinal study: Psychiatric Research Interview for Substance and Mental Disorders, adapted for assessing addiction to opioid analgesics (PRISM-5-OP) | Change from baseline at one year
  Estimation of the incidence of addiction associated with long-term use of opioids for chronic pain.
Cross sectional Study: Prescription Opioid Misuse and Abuse Questionnaire (POMAQ) | Day 1 Assessment
  Estimation of the prevalence of misuse and abuse associated with long term use of opioids for chronic pain.
Cross sectional Study: Psychiatric Research Interview for Substance and Mental Disorders, adapted for assessing addiction to opioid analgesics (PRISM-5-OP) | Day 1 Assessment
  Estimation of the prevalence of addiction associated with long term use of opioids for chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Petronis, Study Chair — Epi Ideas LLC
Locations (2):
- United States (2):
  - Kaiser Permanente Northwest, Portland, Oregon
  - Kaiser Permanente Washington, Seattle, Washington